CLINICAL TRIAL: NCT00719927
Title: Comadres Weight Loss Pilot Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Miriam Hospital (Other)
Responsible Party: Rena Wing, Weight Control and Diabetes Research Center, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2040-08
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2008-06

CONDITIONS: Obesity
Keywords: Social Support
MeSH Terms: conditions — Obesity

ARMS (2):
- 1 (Experimental): Comadre Treatment
  Interventions: Behavioral: Comadres Weight Loss Pilot Program
- 2 (Active Comparator): Non Support Partner Treatment
  Interventions: Behavioral: Comadres Weight Loss Pilot Program

INTERVENTIONS:
Behavioral: Comadres Weight Loss Pilot Program — The first condition will consist of women participating with a female friend (comadre), while the second condition will consist of women participating without a support partner.
  Other Names: Support Partner; Non Support Partner

SUMMARY:
Latinas are more likely to be obese and physically inactive than white women. Therefore, a behavioral weight loss program for Latinas will be tested in this pilot study. Thirty overweight or obese Latinas will be recruited for a 12 week weight loss program at the Weight Control & Diabetes Research Center. Participants will be provided with nutrition and physical activity education and be taught behavioral skills to help them adopt lifestyle changes that produce weight loss. Participants will be placed on a reduced calorie diet and instructed to gradually increase their level of physical activity. To encourage participants to monitor their daily eating and exercise activities, participants will be instructed to record these activities in food and exercise diaries and submit them each week. Two treatment groups will be tested. The first group will have participants attend sessions with a female friend (comadre). The second group will have participants attend sessions without a comadre. The aims of this study are to determine whether we can succeed in recruiting Latinas with their comadres and whether we can reduce participant drop-out by having Latinas participate with their comadres in a behavioral weight loss program.

DETAILED DESCRIPTION:
National studies indicate a need for behavioral treatments for Latinas that promote recommended weight loss and weight loss maintenance practices. In the national Behavioral Risk Factor Surveillance System survey, Latinas were found to be more likely to attempt weight loss than white or black females. However, they were least likely to follow the recommendations of consuming less calories and exercising at least 150 minutes per week. In fact, Latinas more than whites reported using fasting or diet pills as a method of weight control. Furthermore, participating in organized weight loss programs was less common among Latinas than whites. Hence, a weight control intervention aimed at helping Latinas develop the behavioral skills shown to promote weight loss and weight loss maintenance is warranted. We propose to recruit 30 overweight or obese adult Latinas and randomly assign them to one of two conditions. Both conditions will offer 12 weekly group sessions involving a standard behavioral treatment. Behavioral techniques will be taught for the promotion of weight loss via adherence to a reduced caloric diet and increased physical activity. The first condition will consist of women participating with a female friend (comadre), while the second condition will consist of women participating without a support partner. An intervention strategy in which women participate in a behavioral weight loss program with a comadre will be evaluated in terms of participant recruitment and retention in this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Women who self-identify as Hispanic or Latino
* Rhode Island resident
* Overweight or obese (BMI 27-50 kg/m2)
* Ages 18-65 years old
* English speaking & literate
* If randomized to the comadre condition, the participant's comadre must also meet all inclusion and exclusion criteria and must not reside in the same household.

Exclusion Criteria:

* Pregnant, lactating, less than 6 months post-partum, or plans to become pregnant in the next 6 months
* Currently participating in another weight loss program, taking weight loss medication, and/or lost ≥ 10% of body weight during the past 6 months
* Reports being unable to walk 2 blocks (1/4 mile) without stopping
* Reports a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q) (Thomas, Reading, & Shepard, 1992), which will be administered during the phone screen.
* Individuals with medical conditions that could limit exercise will be required to obtain written physician consent to participate
* Reports conditions that in the judgment of the Principal Investigator would render them potentially unlikely to follow the protocol for the study period including terminal illness, plans to relocate, substance abuse, eating disorder, or significant psychiatric problems

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Participant Recruitment and Retention | Sept 2008-March 2009

CONTACTS AND LOCATIONS:
Overall Officials: Rena Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control and Diabetes Research Center, The Miriam Hospital, Providence, Rhode Island, United States